CLINICAL TRIAL: NCT06021210
Title: Letermovir for the Prevention of Cytomegalovirus Infection in Hematopoietic Cell Transplant Recipients Based on the Outcome of Metagenomic Next-Generation Sequencing: a Phase 2, Open Label, Single-Arm Clinical Trial.
Brief Title: Letermovir for the Prevention of CMV Infection in HSCT Recipients Based on the Outcome of mNGS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Xiaowen Tang, The First Affiliated Hospital of Soochow University, The First Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: mNGS+LMV
Record Dates: First submitted 2023-08-26; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: CMV Infection; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — letermovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mNGS detection before stem cell transplantation (Experimental): Using letermovir to prevent CMV reactivation for high-risk patients with pre-existing CMV viremia based on the mNGS detection technology before HSCT
  Interventions: Drug: Letermovir Pill

INTERVENTIONS:
Drug: Letermovir Pill — Letermovir is the world's first and only new drug approved for the prevention of CMV infection. In 2017, it was approved by the U.S. Food and Drug Administration (FDA) for the prevention of CMV infection and disease in CMV-seropositive adult recipients (R+) of allogeneic hematopoietic stem cell transplantation (allo-HSCT). It was approved in China on December 31, 2021.
  Other Names: Letermovir Tablets

SUMMARY:
Letermovir for the Prevention of CMV Infection in HSCT Recipients Based on the Outcome of mNGS

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is widely used as the sole curative treatment for malignant hematological diseases. However, the chances of contracting various pathogenic bacterial infections significantly increase after transplantation, with cytomegalovirus (CMV) infection being the most prevalent [1]. The propotion of CMV-seropositive people ranges from 30% to 97%. After a previous infection, CMV can remain latent in the patient's body and reactivate when the immune function is low, which is the primary cause of CMV infection in allo-HSCT patients, leading to CMV viremia and CMV disease. If CMV viremia progresses to CMV disease, it can invade various organs such as the lungs, digestive tract, retina, and brain, with CMV pneumonia having a mortality rate of over 80% [2]. After allo-HSCT, the incidence of CMV disease ranges from 60% to 70%, depending on the serological status of the donor and recipient [3-4].

In the past, antiviral drugs including ganciclovir, foscarnet, cidofovir, and valganciclovir/valacyclovir were commonly used to treat or prevent CMV infections in clinical practice. These drugs target on viral DNA polymerase, which in turn inhibits the replication of CMV DNA. However, these drugs have serious side effects, such as bone marrow suppression and severe nephrotoxicity, which limit their clinical application.

Letermovir is the world's first and only new drug approved for the prevention of CMV infection. In 2017, it was approved by the U.S. Food and Drug Administration (FDA) for the prevention of CMV infection and disease in CMV-seropositive adult recipients (R+) of allogeneic hematopoietic stem cell transplantation (allo-HSCT). It was approved in China on December 31, 2021. Letermovir targets on the CMV DNA terminase complex consisting of pUL51, pUL56, and pUL89, which affects the formation of appropriate unit-length genomes and interferes with the maturation of virus particles. Therefore, due to its unique pharmacological mechanism, Letermovir does not affect the normal function of human cells, which can avoid the common side effects of other anti-CMV drugs, and it does not develop cross-resistance with other antiviral drugs. Letermovir does not affect the incidence and timing of hematopoietic stem cell implantation and is an effective and safe first-line drug for the prevention of CMV infection and disease after allo-HSCT. It is recommended for CMV-seropositive adult allo-HSCT recipients to use Letermovir for CMV prophylaxis from day 0 after transplantation, no later than day 28 after transplantation (can be used before implantation), and continue until day 100 after transplantation.

The mNGS (metagenomic next-generation sequencing) detection method is a new high-throughput sequencing method for analyzing the microbiome in clinical samples, independent of traditional microbial cultivation. It involves extracting nucleic acid sequences from the samples, constructing sequencing libraries, sequencing the nucleic acid sequences in the sample, and comparing them to a microbial-specific database for analysis. Through intelligent algorithms, it identifies the species information of suspected pathogenic microorganisms with high sensitivity. The mNGS method can detect potential CMV infection in patients before having positive outcomes in qPCR detection of CMV-DNA, and has been used clinically.

This study will evaluate the efficacy and safety of using letermovir to prevent CMV reactivation for high-risk patients with pre-existing CMV viremia based on the mNGS detection technology before HSCT.

ELIGIBILITY:
Inclusion Criteria:

* HSCT candidate who has decided to primary transplant and is willing to participate in the study.
* HSCT candidate undergo mNGS detection before transplantation.

Exclusion Criteria:

* Patients below 14 years ago or above 65 years ago.
* Patients having active infection at the time of letermovir initiation.
* Patient recruited in a clinical study on an anti-CMV trial, or took similar anti-CMV drugs previously.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of clinically significant CMV infection with letermovir prevention after HSCT Defined as CMV DNAemia leading to preemptive treatment or presence of CMV disease | Time from registration to event, max 24 weeks
  The diagnosis of CMV infection is based on CMV-DNA detection of qPCR.

SECONDARY OUTCOMES:
Cumulative incidences of CMV reactivation | Time from registration to event, max 24 weeks
  The cumulative incidences of CMV reactivation after transplantion.
Incidence of Acute and/or chronic graft versus host disease(a/cGVHD) | Time from registration to event, max 24 weeks
  The diagnosis and grading of aGVHD are based on the modified Glucksberg grading standard.
Incidence of transplantation Complications after transplantation | Time from registration to event, max 24 weeks
  Incidence of transplantation Complications such as mucositis, hepatic veno-occlusive disease(SOS), thrombotic microangiopathy(TMA), interstitial pneumonia, hemorrhagic cystitis, infections etc.
Incidence of CMV-related disease mortality | Time from registration to event, max 24 weeks
  The Incidence of CMV-related disease mortality after transplantation.
Incidence of all-cause mortality and non-relapse mortality | Time from registration to event, max 24 weeks
  The Incidence of all-cause mortality and non-relapse mortality after transplantion.
Leukemia-free survival(LFS) | Time from registration to event, max 24 weeks
  Leukemia-free survival(LFS) is defined as the time from enrollment to relapse of primary disease or death from any cause.
Overall survival(OS) | Time from registration to event, max 24 weeks
  Overall survival(OS) is defined as the time from transplantation to death resulting from any cause.
GVHD-free and relapse-free survival(GRFS) | Time from registration to event, max 24 weeks
  GRFS is defined as the time from graft infusion to the onset of grades 3 to 4 aGVHD, moderate to severe cGVHD, or relapse/disease progression/death.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowen Tang, PhD, Study Chair — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No